CLINICAL TRIAL: NCT06025890
Title: Early Clinical Evaluation and Intervention of Developmental Behavioral Diseases Based on Multicenter Cohort Study
Brief Title: Clinical Evaluation and Intervention of Developmental Behavioral Diseases Based on Multicenter Cohort Study(CEIDBDBMCS)
Acronym: CEIDBDBMCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Li (Other)
Collaborators: Southeast University, China (Other); East China Normal University (Unknown); Shanghai Children's Medical Center (Other); Seventh Medical Center of PLA Army General Hospital (Other)
Responsible Party: Sponsor-Investigator, Chen Li, Associate Professor, Director, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CEIDBDBMCS
Record Dates: First submitted 2023-01-31; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: ADHD; Language Disorders
Keywords: ADHD; Language Disorder; Artificial Intelligence; fNIRS
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Language Disorders

STUDY DESIGN:
Intervention Model Description: Collect blood samples from 600 cases of language disorder and 800 cases of ADHD, and complete an fNIRS task test from 800 ADHD patients. Based on the modularization of "core ability improvement", "specific ability improvement and ability strategy acquisition", "learning problems and interpersonal relationships", "social adaptation"; and other programs, sometimes combined with computer-aided cognitive training, parenting behavior management training, and/or mindfulness training, aerobic exercise, and other intervention forms can achieve personalized functional training intervention for children. Use brain near-infrared imaging technology to capture multimodal neuroimaging features of young children; use high-precision repetitive transcranial direct current stimulation technology to conduct positive neural enhancement and adjustment training on the target brain area.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Language Disorder (Experimental): The language disorder group had to complete a two-year follow-up and intervention. Collect blood samples from 600 cases of language disorder.
  Interventions: Other: Functional Training.; Other: Observe.
- Attention Deficit Hyperactivity Disorder (Experimental): The ADHD group had to complete a two-year follow-up and intervention.Collect blood samples 800 cases of ADHD, and complete a fNIRS task test from 800 ADHD patients.
  Interventions: Other: Functional Training.; Other: Observe.
- Normal children (No Intervention): For children aged 1-4, 2 developmental behavioral specialists with associate professor titles or above exclude language barriers.
- Healthy children (No Intervention): Children aged 3-6, except ADHD with 2 developmental behavioral and/or psychiatrists with associate professor titles or above.

INTERVENTIONS:
Other: Functional Training. — Based on the modularization of "core ability improvement", "specific ability improvement and ability strategy acquisition", "learning problems and interpersonal relationships", "social adaptation"; and other programs, sometimes combined with computer-aided cognitive training, parenting behavior management training and/or mindfulness training, aerobic exercise and other intervention forms, can achieve personalized functional training intervention for children. Use brain near-infrared imaging technology to capture multimodal neuroimaging features of young children; use high-precision repetitive transcranial direct current stimulation technology to conduct positive neural enhancement and adjustment training on the target brain area. Based on physical therapy stimulation, neuromodulation improves core symptoms in children.
  Arms: Attention Deficit Hyperactivity Disorder; Language Disorder
Other: Observe. — Children with language disorders and ADHD were recruited at an early age when symptoms first appeared. Professional assessments were conducted to evaluate clinically relevant developmental and cranial nerve function indicators using near-infrared brain imaging technology. Follow-up was conducted for two years, and the outcome indicators were language disorder and attention deficit hyperactivity disorder.
  Arms: Attention Deficit Hyperactivity Disorder; Language Disorder

SUMMARY:
Diagnosis of Language Disorder and Attention Deficit Hyperactivity Disorder (ADHD) is difficult for several reasons. This study aims to establish a Chinese multi-center cohort for the early diagnosis of language disorder and ADHD in children, develop appropriate early assessment tools and formulate intervention programs and standards for early functional training. Based on a national multi-center research team with Chongqing, Shanghai, and Beijing as the core areas, the investigators established a specific disease cohort for early diagnosis of language disorder and ADHD: a specific disease cohort with language disorder (900 cases) who were 1-3 years when the follow-up started, and 4-6 years old at the end of follow-up; a specific cohort with ADHD (1200 cases) who were 3-6 years when the follow-up started, and 7-9 years old at the end of follow-up. At the time of enrollment, professional assessments such as clinical development indicators and neurological function indicators were assessed using functional near-infrared spectroscopy(fNIRS). Outcome measures were speech impairment and hyperactivity. Blood samples were taken from 600 speech-impaired patients and 800 ADHD patients. Of these, 800 ADHD subjects completed an fNIRS imaging task. Build an intelligent brain image big data analysis system to realize early quality control, processing, and analysis of brain images, and study objective markers for early disease detection. The investigators can use machine learning and applications for early diagnosis, developing big data analysis tools such as integrated clinical assessment and brain imaging, promoting comprehensive clinical assessment and big data analysis tools systems such as brain imaging, and building assessment tools for language disorders and ADHD. Through the implementation and results of the multi-center special disease cohort platform, evidence-based medical evidence is collected to form clinical standards and guidelines.

DETAILED DESCRIPTION:
1. Procedures. From December 2022 to May 2024, the research team completed the collection and follow-up of 900 cases of language disorder and 1,200 cases of ADHD, and included them in the language disorder and ADHD cohort case collection database.From June 2024 to November 2024, 900 children with language disorders and 1,200 children with ADHD will be followed; blood samples will be collected from 600 children with language disorders and 800 children with ADHD; 800 children with ADHD will be completed using the fNIRS task test. From December 2024 to November 2025, complete the follow-up of 900 cases of language disorder and 1,200 cases of ADHD, complete the development of an early assessment tool set suitable for the Chinese children with language disorders and ADHD, complete the formulation of intervention plans, establish a unified standard, and extended the results to 50 hospitals.
2. Sample size. This study is an intervention study. The language disorder group and the ADHD group had to complete a two-year follow-up and intervention. collect blood samples from 900 cases of language disorder and 1,200 cases of ADHD, and complete an fNIRS task test from 800 ADHD patients. The primary endpoints were language disorder and ADHD.An electronic data acquisition system with a follow-up management module, multi-level authority management and automatic SMS notification function is adopted to build an integrated and standardized multi-center queue data storage and sharing platform. Based on the modularization of "core ability improvement", "specific ability improvement and ability strategy acquisition", "learning problems and interpersonal relationships", "social adaptation"; and other programs, sometimes combined with computer-aided cognitive training, parenting behavior management training and/or mindfulness training, aerobic exercise and other intervention forms can achieve personalized functional training intervention for children. Use brain near-infrared imaging technology to capture multimodal neuroimaging features of young children; use high-precision repetitive transcranial direct current stimulation technology to conduct positive neural enhancement and adjustment training on the target brain area. Based on physical therapy stimulation, neuromodulation improves core symptoms in children.
3. Statistical analysis. By integrating multiple methods such as scale evaluation, behavioral testing, and experience sampling into the tool library, digitization, and interface visualization are realized. Combined with the multi-center cloud data platform, a generalized linear probability model is created, and an early evaluation tool is established. Capturing multimodal neuroimaging features of early childhood using fNIRS; training a hierarchical machine learning scoring model using fused neural features. Based on the classic support vector machine algorithm, the detection model is trained with the post-diagnosis as the result label, and the leave-one-out cross-validation method is used for testing.
4. Ethical matters and data protection. The patients who participated in the study will sign the informed consent (obtained from the guardian). And this study was approved by the local ethics committee. The patient's name will be abbreviated and the research data will be assigned a code then to provide to the researcher. The authorization from parents on the patient's health information remains valid until the study is completed. After that, researchers will delete private information from the study record.

ELIGIBILITY:
1. Language disorder

Inclusion criteria:

1. Language disorder(n=900): This study included children between the ages of 1-4 who were evaluated for potential language disorder by two developmental behavioral specialists holding the title of associate professor or higher.
2. Control group(n=100): This study included children between the ages of 1-4 who were exclude with language disorder by two developmental behavioral specialists with the title of associate professor or higher.

Exclusion criteria:

1. Children with a history of language development delay or language disorder intervention treatment.
2. DQ score below 85.
3. (3) Patients with organic diseases of the nervous system, epilepsy, autism spectrum disorder, global developmental delay, and hearing impairment, and/or people caring for patients with mental illness, hearing impairment,language disoeder.

2.ADHD

Inclusion criteria:

1. ADHD(n=1200): This study included children between the ages of 3-6 who were evaluated for potential ADHD by two developmental behavioral and/or psychiatrists with the rank of associate professor or higher.
2. Control group(n=100):This study included children between the ages of 1-4 who were exclude with ADHD by two developmental behavioral and/or psychiatrists with the rank of associate professor or higher.

Exclusion criteria:

1. Children with ADHD intervention treatment.
2. DQ score lower than 85, or IQ score lower than 80.
3. Patients with organic diseases of the nervous system, epilepsy, autism spectrum disorder, global developmental delay, mental retardation, atopic dermatitis, asthma, hearing impairment or visual impairment.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2100 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Changes in the Gesell Developmental Scale(GDS). | 2 years
  Children are followed up every 6 months, and at each follow-up point, the GDS is used to assess children and obtain their comprehensive scores in various developmental domains. These domains may include motor development, gross and fine motor coordination, language and communication, cognitive and thinking abilities. The score range for language development is 0-100, where a higher score indicates a more excellent level of development in the field, in line with age expectations, while a lower score may indicate a lag or issues in the development of that field.
Changes in Infants-Junior High School Students'Social Development Screening Test. | 2 years
  The scores obtained from the Infant to Middle School Student Social Life Skills Scale (S-M) at each 3-month follow-up reflect the social interaction, communication skills, and adaptation to social environments of the participants at different follow-up stages. The score range for the Infants-Junior High School Students' Social Development Screening Test varies depending on the specific assessment tool used. Generally, the scores may range from 0 to 100 or may be presented in percentile ranks. In general, a higher score indicates that the individual's social development is more advanced and aligned with age expectations. On the other hand, a lower score might suggest developmental lags or challenges in social skills.
Changes in Dream-Infant-Toddler Language Communication Screening（DREAM-IT-S） | 2 years
  The scores obtained from the Dream-Infant-Toddler Language Communication Screening (DREAM-IT-S) administered at each 3-month follow-up reflect the language abilities of children.The total score range of DREAM-IT-S is between 0 and 10, where a lower score indicates better language communication ability, while a higher score suggests potential delays or obstacles in language development.
Changes in Dreaming Children's Language Standardized Assessment (DREAM-C) | 2 years
  The scores obtained from the Dream-Infant-Toddler Language Communication Screening (DREAM-IT-S) and Dreaming Children's Language Standardized Assessment (DREAM-C) administered at each 3-month follow-up reflect the language abilities of children. The total score range of DREAM-C can vary depending on the specific assessment criteria, but it typically falls within a predetermined range. The exact range depends on the design of the assessment tool and scoring system, but generally, it may be scored on a scale from 0 to 100 or other values. Lower scores indicate stronger language abilities and effective communication skills, while higher scores may suggest potential language development delays or communication barriers.
Changes in Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) . | 2 years
  Conducting follow-up assessments every 6 months using the Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) scores reflect the cognitive and intellectual development of children at different follow-up points. The total score range of WPPSI-IV is in percentage (from 0 to 100), where higher scores indicate stronger abilities in the corresponding domains.
Changes in Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV). | 2 years
  Conducting follow-up assessments every 6 months using the Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) scores reflect the cognitive and intellectual development of children at different follow-up points. The total score range of WISC-IV is in percentage (from 0 to 100), where higher scores indicate stronger abilities in the corresponding domains.
Changes in Child Behavior Checklist (CBCL) | 2 years
  Conducting follow-up assessments every 3 months using the Child Behavior Checklist (CBCL) scores reflects the emotional and behavioral issues of children at different follow-up points.The scores on the CBCL typically range from 0 to 100, and higher scores may indicate that children are experiencing difficulties in behavior and emotional problems.
Changes in the Vanderbilt Assessment Scale | 2 yaers
  The use of the Vanderbilt Assessment Scale scores in follow-up visits every three months reflects the ADHD symptomatology of children at different follow-up milestones. The total score of the Vanderbilt Assessment Scale can range from 0 to 54. A higher score indicates a greater likelihood of ADHD symptoms or difficulties with attention and behavior.
Changes in Questionnaire-Children with Difficulties. | 2 years
  Follow-up assessments every 3 months, using the Questionnaire-Children with Difficulties (QCD) scores, reflect children's psychological issues and behavioral difficulties. The scoring range of the QCD questionnaire may vary depending on the specific version or rating system. For example, certain rating systems may categorize scores into levels of severity such as mild, moderate, or severe difficulties. Higher scores may indicate higher levels of psychological difficulties or disorders. Conversely, lower scores may suggest fewer problems or mild manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, doctor, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Growth, Development and Mental health of Children and Adolescence Center, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.

REFERENCES:
- [Background] Wolraich ML, Bard DE, Neas B, Doffing M, Beck L. The psychometric properties of the Vanderbilt attention-deficit hyperactivity disorder diagnostic teacher rating scale in a community population. J Dev Behav Pediatr. 2013 Feb;34(2):83-93. doi: 10.1097/DBP.0b013e31827d55c3. PMID 23363973
- [Background] Elvsashagen T, Shadrin A, Frei O, van der Meer D, Bahrami S, Kumar VJ, Smeland O, Westlye LT, Andreassen OA, Kaufmann T. The genetic architecture of the human thalamus and its overlap with ten common brain disorders. Nat Commun. 2021 May 18;12(1):2909. doi: 10.1038/s41467-021-23175-z. PMID 34006833
- [Background] Kim JH, Kim JY, Lee J, Jeong GH, Lee E, Lee S, Lee KH, Kronbichler A, Stubbs B, Solmi M, Koyanagi A, Hong SH, Dragioti E, Jacob L, Brunoni AR, Carvalho AF, Radua J, Thompson T, Smith L, Oh H, Yang L, Grabovac I, Schuch F, Fornaro M, Stickley A, Rais TB, Salazar de Pablo G, Shin JI, Fusar-Poli P. Environmental risk factors, protective factors, and peripheral biomarkers for ADHD: an umbrella review. Lancet Psychiatry. 2020 Nov;7(11):955-970. doi: 10.1016/S2215-0366(20)30312-6. PMID 33069318
- [Background] Chang JP, Su KP, Mondelli V, Pariante CM. Omega-3 Polyunsaturated Fatty Acids in Youths with Attention Deficit Hyperactivity Disorder: a Systematic Review and Meta-Analysis of Clinical Trials and Biological Studies. Neuropsychopharmacology. 2018 Feb;43(3):534-545. doi: 10.1038/npp.2017.160. Epub 2017 Jul 25. PMID 28741625
- [Background] Zhao J, Yu Z, Sun X, Wu S, Zhang J, Zhang D, Zhang Y, Jiang F. Association Between Screen Time Trajectory and Early Childhood Development in Children in China. JAMA Pediatr. 2022 Aug 1;176(8):768-775. doi: 10.1001/jamapediatrics.2022.1630. PMID 35666518